CLINICAL TRIAL: NCT05750589
Title: Randomized, Controlled, Double-Masked Study to Evaluate the Efficacy of IRX-101 in Reducing Post-Intravitreal Pain and Corneal Epitheliopathy
Brief Title: Safety and Tolerability of IRX-101 in Patients Receiving Intravitreal Injections
Acronym: COMFORT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: iRenix Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRX-2022-001
Record Dates: First submitted 2023-02-17; First posted 2023-03-01 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Retinal Disease
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to IRX-101 or Providone-Iodine
Who Masked: Participant, Investigator
Masking Description: Treatment assignment will be unknown (or masked) to the study subjects, the evaluating physician, the Sponsor and its agents (with the exception of personnel performing randomization, unmasked drug accountability study monitors, and corporate compliance staff). The treating physician will be unmasked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IRX-101 (Experimental): Subjects randomized to IRX-101 will receive the investigational product, IRX-101.
  Interventions: Drug: IRX-101
- 5% Povidone-iodine (Active Comparator): Subjects randomized to this arm will receive the standard of care, Providone-iodine, at a concentration of 5%.
  Interventions: Drug: Providone-Iodine

INTERVENTIONS:
Drug: IRX-101 — IRX-101 is a novel ocular anti-septic
  Arms: IRX-101
Drug: Providone-Iodine — 5% Providone-Iodine
  Arms: 5% Povidone-iodine

SUMMARY:
This is a randomized, double-masked study to evaluate the tolerability and safety of IRX-101 versus 5% povidone-iodine (PI) in subjects receiving intravitreal anti-VEGF injections.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving informed consent
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, ≥ 18 years of age and receiving intravitreal anti-VEGF injections in one or both eyes

Exclusion Criteria:

1. Current or past diagnosis of endophthalmitis
2. Current diagnosis of uveitis
3. Monocular patients (vision 20/100 or worse in one eye) who are receiving injections in the better seeing eye
4. Current use of viscous lidocaine products for ocular anesthesia prior to IVT
5. Currently receiving intravitreal steroid injections
6. Concurrent participation in another clinical trial
7. Females who are pregnant, planning to become pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of post-intravitreal injection eye pain | Demonstrate a reduction in mean 1-hr post-injection pain scores
  Demonstrate the superiority of IRX-101 compared to PI in terms of reducing patient-reported post-intravitreal injection eye pain; pain will be assessed using the visual analog pain scale, a validated patient-reported outcome measure (questionnaire) for assessing patient's subjective pain and discomfort

SECONDARY OUTCOMES:
Change in post-IVT corneal epitheliopathy as evaluated by corneal fluorescein staining scores | Immediately following intraviteral injection
  Demonstrate the superiority of IRX-101 compared to PI in terms of reducing corneal epitheliopathy / corneal fluorescein staining post-intravitreal injection; corneal staining will be obtained using validated Oxford Corneal Staining scale of 0 (no staining) to 5 (maximal corneal staining)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Smith, MD, Study Chair — Founder
Locations (1):
- R. Gary Lane, II MD, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided